CLINICAL TRIAL: NCT01026402
Title: A Phase I, Open Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the mTor Kinase Inhibitor AZD2014 Administered Orally to Patients With Advanced Solid Malignancies
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Preliminary Efficacy of AZD2014
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2270C00001; 2009-015244-42 (EudraCT Number)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Advanced Solid Malignancies
Keywords: Phase I; cancer; advanced solid malignancies; dose escalation; AZD2014; mTor kinase inhibitor; safety; pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD2014 (Experimental): AZD2014 dose escalation phase in Part A and expansion phase in Part B.
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014 — Dose escalation phase: a single dose taken orally (solution or tablet) of AZD2014 on single dose day 1 (visit 2), followed by once or twice daily continuous dosing after a washout period (48 hours - 7 days) at visit 4, until discontinuation or withdrawal or Single or multiple doses taken orally (solution or tablet) of AZD2014 taken intermittently until discontinuation or withdrawal. Expansion phase: twice daily dosing from day 1 until discontinuation or withdrawal or a single dose taken orally of AZD2014 on single dose day 1 (visit 2), followed by a single dose on second single dose day 1 (visit 3) after a washout period (48 hours - 7 days) followed by once or twice daily continuous dosing after a washout period (48 hours - 7 days) at visit 4, until discontinuation or withdrawal or single or multiple doses taken orally (solution or tablet) of AZD2014 taken intermittently until discontinuation or withdrawal.

SUMMARY:
The main purpose of the study is to establish a safe dose of the drug by providing information on any potential side effects this drug may cause and collecting data about how a patient's cancer responds to the drug. The study will also assess the blood levels and action of AZD2014 in the body over a period of time and will indicate whether the drug has an effect on the types of cancer the patients have.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of a solid, malignant tumour that is refractory to standard therapies or for which no standard therapies exist
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by computerised tomography (CT) magnetic resonance imaging (MRI) or plain X-ray and is suitable for repeated assessment
* World Health Organisation performance status 0-2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks

Exclusion Criteria:

* Patients with severe laboratory abnormalities for haematology, liver or renal function. Also treatment with any haemopoietic growth factors are not allowed within two weeks prior to first dose of study drug
* Patients with abnormal fasting glucose, type I or uncontrolled type II diabetes
* Patients with severe cardiac condition of ischemia, impaired ventricular function and arrhythmias, evidence of severe or uncontrolled systemic or current unstable or uncompensated respiratory or cardiac conditions

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Udai Banerji, Principal Investigator — The Royal Marsden NHS Foundation Trust, Downs Road, Sutton, Surrey SM2 5PT; Elisabeth Oelmann, Study Director — AstraZeneca
Locations (2):
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject In: 30th December 2009 Last Subject Last visit: 18th August 2014 2 sites located in the UK Number of participants analyzed in Dose Limiting Toxicity (DLT) outcome measure are patients evaluable for DLT assessment Note - in the Clinical Study Report, combined groups are discussed (e.g. Part A 125mg BD Int and Part B 125mg BD tab Int)
Pre-assignment Details: A total of 172 patients were enrolled. 135 of these patients passed screening assessments and were dosed
Groups:
- Part A 25mg BD Soln Cont; Part A 50mg BD Soln Cont; Part B 50mg BD Soln Cont; Part B Fed/Fasted 50mg BD Tab Cont; Part A 70mg BD Soln Cont; Part A 100mg BD Soln Cont: Continuous BD dosing
- Part A 75mg QD Soln Cont; Part A 125mg QD Soln Cont; Part A 100mg QD Tab Cont; Part A 125mg QD Tab Cont; Part A 175mg QD Tab Cont: Continuous QD dosing
- Part A 100mg BD Tab Int; Part A 125mg BD Tab Int; Part A 170mg BD Tab Int; Part A 225mg BD Tab Int; Part B 125mg BD Tab Int; Part B 170mg BD Tab Int: Intermittent BD dosing
Period: Overall Study
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Started | 6 | 8 | 33 | 18 | 3 | 5 | 8 | 3 | 7 | 3 | 7 | 8 | 8 | 6 | 3 | 5 | 4
Completed | 6 | 8 | 33 | 18 | 3 | 5 | 8 | 3 | 7 | 3 | 7 | 8 | 8 | 6 | 3 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set - All patients that received at least 1 dose of AZD2014. This includes dosed patients who are not evaluable for dose escalation decision purposes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Total
Number analyzed (Participants) | 6 | 8 | 33 | 18 | 3 | 5 | 8 | 3 | 7 | 3 | 7 | 8 | 8 | 6 | 3 | 5 | 4 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (15.8) | 58.3 (14.1) | 57.2 (10.3) | 58.6 (14.2) | 51.7 (11.5) | 50.0 (16.1) | 59.4 (11.0) | 51.3 (18.9) | 65.6 (9.8) | 59.0 (18.7) | 67.3 (7.9) | 57.6 (5.4) | 53.8 (9.9) | 54.2 (14.2) | 42.7 (9.0) | 47.4 (14.8) | 50.0 (8.2) | 56.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 22 | 8 | 2 | 4 | 6 | 2 | 4 | 3 | 4 | 4 | 6 | 5 | 3 | 3 | 2 | 88
  Male | 4 | 0 | 11 | 10 | 1 | 1 | 2 | 1 | 3 | 0 | 3 | 4 | 2 | 1 | 0 | 2 | 2 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Maximum Tolerated Dose (MTD) was determined by testing various doses and schedules of AZD2014 in cohorts of 3-6 evaluable patients. MTD reflects the highest dose of drug at each schedule that did not cause a DLT in >1 patient
Time Frame: Up to 21 days from first multiple dose
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 6 | 6 | 0 | 0 | 3 | 3 | 6 | 2 | 2 | 3 | 6 | 6 | 5 | 6 | 3 | 4 | 4
Participants | 0 | 0 |  |  | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 4
Statistical Analysis 1: Comparison: Part A 25mg BD Soln Cont vs Part A 50mg BD Soln Cont vs Part A 70mg BD Soln Cont vs Part A 100mg BD Soln Cont; Test type: Superiority or Other; Maximum Tolerated Dose = 50 — 50mg twice daily continuous dosing 20 evaluable patients
Statistical Analysis 2: Comparison: Part A 75mg QD Soln Cont vs Part A 125mg QD Soln Cont vs Part A 100mg QD Tab Cont vs Part A 125mg QD Tab Cont vs Part A 175mg QD Tab Cont; Test type: Superiority or Other; Maximum Tolerated Dose = 100 — 100mg once daily continuous dosing 16 evaluable patients
Statistical Analysis 3: Comparison: Part A 100mg BD Tab Int vs Part A 125mg BD Tab Int vs Part A 170mg BD Tab Int vs Part A 225mg BD Tab Int vs Part B 125mg BD Tab Int vs Part B 170mg BD Tab Int; Test type: Superiority or Other; Maximum Tolerated Dose = 125 — 125mg twice daily intermittent dosing (2 days on, 5 days off) 29 evaluable patients

2. Secondary Outcome: Best Objective Response
Description: Best Objective Response per Response Evaluation Criteria in Solid Tumours Criteria (RECIST) 1.1 for target and non target lesions assessed by CT, MRI or X-ray; Complete Response (CR), Disappearance of all target lesions since baseline; Partial Response (PR), At least a 30 percent decrease in the sum of diameters of target lesions; Progressive Disease (PD), At least a 20 percent increase in the sum of diameters of target lesions and an absolute increase of at least 5mm
Time Frame: Assessed every 8 weeks until progression or withdrawal, whichever came first, estimated to be up to 4 months
Population: Efficacy analysis set - Patients who received at least 1 dose of AZD2014 and have a baseline tumour assessment
Measure: Number; unit: Participants
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 6 | 8 | 33 | 18 | 3 | 5 | 8 | 3 | 7 | 3 | 7 | 8 | 8 | 6 | 3 | 5 | 4
Participants
  Responders | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Non-responders | 6 | 8 | 31 | 18 | 3 | 5 | 8 | 3 | 7 | 3 | 7 | 8 | 8 | 6 | 3 | 5 | 4
  Stable disease ≥8 wks (a subset of non-responders) | 2 | 1 | 12 | 7 | 1 | 1 | 4 | 0 | 1 | 0 | 3 | 2 | 1 | 1 | 0 | 2 | 0

3. Secondary Outcome: Maximum Concentration (Cmax) Single Dose
Description: Maximum concentration following single dose (n varies between PK outcome measures as a subset of the PK analysis set was used with reportable AZD2014 plasma concentrations and PK parameters at that visit who have no important adverse events or protocol deviations that may impact PK at that visit, which means that different amounts of data were available for different parameters depending on what visits the parameter covered)
Time Frame: Following Single Dose up to 12, 24 or 48 hours post dose
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B 50mg BD Tablet Fasted; Part B 50mg BD Tablet Fed: Continuous BD dosing
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 6 | 8 | 19 | 0 | 3 | 4 | 8 | 3 | 7 | 3 | 7 | 8 | 8 | 6 | 3 | 5 | 4 | 18 | 18
ng/mL | 435 (41.98) | 1313 (43.62) | 1089 (62.43) |  | 1476 (78.18) | 4046 (22.46) | 2048 (47.26) | 2989 (20.69) | 3251 (54.69) | 1868 (32.82) | 1826 (62.99) | 3293 (74.44) | 5223 (39.53) | 2849 (61.7) | 4395 (14.92) | 2382 (38.8) | 2787 (71.97) | 856.3 (73.47) | 643.7 (54.10)

4. Secondary Outcome: Area Under the Curve (AUC) Single Dose
Description: Area under the curve following single dose Continuous dosing - AUC parameter used Intermittent dosing - AUC(0-12) used (n varies between PK outcome measures as a subset of the PK analysis set was used with reportable AZD2014 plasma concentrations and PK parameters at that visit who have no important adverse events or protocol deviations that may impact PK at that visit, which means that different amounts of data were available for different parameters depending on what visits the parameter covered)
Time Frame: Following Single Dose up to 12, 24 or 48 hours post dose
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 6 | 8 | 17 | 0 | 3 | 4 | 8 | 3 | 6 | 3 | 7 | 8 | 8 | 6 | 3 | 5 | 4 | 17 | 16
ng*h/mL | 1640 (51.92) | 5308 (63.35) | 3520 (81.37) |  | 8866 (50.78) | 20790 (39.4) | 11160 (64.18) | 23450 (24) | 31670 (61.45) | 11850 (11.29) | 8364 (118.6) | 18630 (74.75) | 33840 (60.95) | 15390 (50.33) | 30030 (14.13) | 8967 (32.54) | 9671 (65.88) | 3690 (98.07) | 3411 (66.71)

5. Secondary Outcome: Maximum Concentration (Cmax) at Steady State
Description: Cmax at steady state (n varies between PK outcome measures as a subset of the PK analysis set was used with reportable AZD2014 plasma concentrations and PK parameters at that visit who have no important adverse events or protocol deviations that may impact PK at that visit, which means that different amounts of data were available for different parameters depending on what visits the parameter covered)
Time Frame: Multiple dosing to steady state (up to 12 or 48 hours post dose)
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 6 | 6 | 11 | 0 | 2 | 3 | 6 | 0 | 0 | 3 | 6 | 6 | 3 | 6 | 1 | 2 | 0 | 14 | 0
ng/mL | 746.9 (72.42) | 1822 (38.78) | 1704 (85.92) |  | NA (NA) — When there were less than 3 values, summary values were not calculated | 5517 (29.14) | 2730 (47.23) |  |  | 3258 (25.20) | 3534 (25.08) | 7557 (38.19) | 11400 (24.23) | 5649 (27.38) | NA (NA) — When there were less than 3 values, summary values were not calculated | NA (NA) — When there were less than 3 values, summary values were not calculated |  | 1162 (46.37) |

6. Secondary Outcome: Area Under the Curve (AUC) at Steady State
Description: AUC at steady state Continuous dosing - AUCss used Intermittent dosing - Weekly AUC used (n varies between PK outcome measures as a subset of the PK analysis set was used with reportable AZD2014 plasma concentrations and PK parameters at that visit who have no important adverse events or protocol deviations that may impact PK at that visit, which means that different amounts of data were available for different parameters depending on what visits the parameter covered)
Time Frame: Multiple dosing to steady state (up to 12 or 48 hours post dose)
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 6 | 6 | 11 | 0 | 1 | 1 | 6 | 0 | 0 | 3 | 6 | 6 | 3 | 5 | 1 | 2 | 0 | 11 | 0
ng*h/mL | 2984 (78.71) | 6436 (57.04) | 7532 (120.5) |  | NA (NA) — When there were less than 3 values, summary values were not calculated | NA (NA) — When there were less than 3 values, summary values were not calculated | 17230 (64.89) |  |  | 77690 (41.93) | 78150 (73.52) | 177100 (79.93) | 380200 (52.06) | 89530 (27.06) | NA (NA) — When there were less than 3 values, summary values were not calculated | NA (NA) — When there were less than 3 values, summary values were not calculated |  | 5275 (53.17) |

7. Secondary Outcome: Urine PK - Fraction Dose Excreted (fe(0-12)) Single Dose
Description: Fraction dose excreted unchanged in the urine from 0-12 hours after a single dose (n varies between PK outcome measures as a subset of the PK analysis set was used with reportable AZD2014 plasma concentrations and PK parameters at that visit who have no important adverse events or protocol deviations that may impact PK at that visit, which means that different amounts of data were available for different parameters depending on what visits the parameter covered)
Time Frame: Pre dose through to 12 hours post dose
Population: PK analysis set - A subset of Safety Analysis set who have reportable plasma concentrations and PK parameter data and who have no important protocol deviations/AEs that may impact PK
Measure: Mean (Standard Deviation); unit: Percent concentration
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 5 | 7 | 0 | 0 | 2 | 4 | 4 | 0 | 6 | 0 | 5 | 6 | 7 | 1 | 1 | 5 | 3 | 0 | 0
Percent concentration | 0.3709 (0.2953) | 0.5459 (0.4828) |  |  | NA (NA) — When there were less than 3 values, summary values were not calculated | 0.7094 (0.3569) | 0.7728 (0.4854) |  | 0.8344 (0.5690) |  | 0.8991 (0.7350) | 0.4744 (0.2252) | 1.106 (0.8091) | NA (NA) — When there were less than 3 values, summary values were not calculated | NA (NA) — When there were less than 3 values, summary values were not calculated | 0.3288 (0.1359) | 0.7680 (0.7217) |  |

8. Secondary Outcome: Urine PK - Fraction Dose Excreted (fe(0-12)) at Steady State
Description: Fraction dose excreted unchanged in the urine from 0-12 hours after dosing (n varies between PK outcome measures as a subset of the PK analysis set was used with reportable AZD2014 plasma concentrations and PK parameters at that visit who have no important adverse events or protocol deviations that may impact PK at that visit, which means that different amounts of data were available for different parameters depending on what visits the parameter covered)
Time Frame: Pre dose through to 24 hours post dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent concentration
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percent concentration |  |  |  |  | NA (NA) — When there were less than 3 values, summary values were not calculated | 0.9056 (0.6456) | 1.026 (0.3658) |  |  |  |  |  |  |  |  |  |  |  |

9. Secondary Outcome: Urine PK - Renal Clearance (Renal CL) Single Dose
Description: Renal Clearance (n varies between PK outcome measures as a subset of the PK analysis set was used with reportable AZD2014 plasma concentrations and PK parameters at that visit who have no important adverse events or protocol deviations that may impact PK at that visit, which means that different amounts of data were available for different parameters depending on what visits the parameter covered)
Time Frame: Pre dose through to 24 hours post dose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 5 | 6 | 0 | 0 | 2 | 4 | 3 | 0 | 5 | 0 | 6 | 6 | 7 | 1 | 1 | 5 | 3 | 0 | 0
L/h | 0.07304 (0.07247) | 0.03994 (0.02933) |  |  | NA (NA) — When there were less than 3 values, summary values were not calculated | 0.04338 (0.009039) | 0.07526 (0.03353) |  | 0.08576 (0.02948) |  | 0.1081 (0.01434) | 0.06049 (0.05774) | 0.07377 (0.05802) | NA (NA) — When there were less than 3 values, summary values were not calculated | NA (NA) — When there were less than 3 values, summary values were not calculated | 0.03083 (0.01394) | 0.09813 (0.04768) |  |

10. Secondary Outcome: Urine PK - Renal Clearance (Renal CL) at Steady State
Description: as for outcome 9
Time Frame: Pre dose through to 24 hours post dose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont | Part B 50mg BD Tablet Fasted | Part B 50mg BD Tablet Fed
Number analyzed (Participants) | 5 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
L/h | 0.03702 (0.02688) | 0.04242 (0.01126) |  |  |  |  |  |  |  |  |  |  |  |  |  | NA (NA) — When there were less than 3 values, summary values were not calculated |  |  |

11. Secondary Outcome: Percent Change From Baseline in p4EBP1 at 2 Hours Post Dose
Description: Phosphorylation levels of 4EBP1 from peripheral blood mononuclear cell (Patients with undetectable values at baseline have been excluded)
Time Frame: predose and 2 hours after a single dose
Population: Efficacy analysis set
Measure: Median (Full Range); unit: Percent change
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 0 | 6 | 13 | 16 | 2 | 5 | 6 | 3 | 7 | 3 | 4 | 7 | 7 | 5 | 2 | 5 | 4
Percent change |  | -47.422 [-94.28 to 37.28] | -31.067 [-96.92 to -10.98] | -21.710 [-89.58 to 33.33] | -78.760 [-87.10 to -70.42] | -74.053 [-96.18 to -66.35] | -66.855 [-99.10 to -52.91] | -68.966 [-88.00 to -19.68] | -82.249 [-88.87 to -49.92] | -57.317 [-90.62 to -38.04] | -76.977 [-87.69 to -8.92] | -67.275 [-88.32 to -15.20] | -55.847 [-90.47 to -46.18] | -42.632 [-55.37 to -16.19] | -64.855 [-91.14 to -38.57] | -57.143 [-94.85 to -34.25] | -62.775 [-89.32 to 20.25]

12. Secondary Outcome: Percent Change From Baseline in pAKT (S473) in Platelet Rich Plasma (PRP) at 2 Hours Post Dose
Description: Phosphorylation levels of AKT from PRP (Patients with undetectable values at baseline have been excluded)
Time Frame: predose and 2 hours after a single dose
Population: Efficacy analysis set
Measure: Median (Full Range); unit: Percent change
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 5 | 8 | 32 | 18 | 3 | 5 | 8 | 3 | 7 | 3 | 5 | 8 | 8 | 3 | 2 | 5 | 4
Percent change | -63.633 [-89.99 to -12.15] | -76.202 [-100.00 to 13.47] | -65.375 [-99.99 to 2.29] | -62.942 [-85.01 to 1.74] | -67.349 [-85.26 to -8.86] | -82.737 [-90.39 to -65.60] | -76.364 [-82.05 to -19.42] | -49.476 [-55.87 to -4.13] | -86.422 [-91.65 to -38.57] | -57.326 [-87.40 to -54.24] | -63.350 [-92.14 to -7.03] | -62.839 [-80.97 to 18.61] | -85.376 [-93.44 to -71.63] | -92.031 [-92.12 to -69.58] | -66.958 [-94.85 to -39.07] | -90.374 [-100.00 to -59.13] | -88.343 [-94.48 to -71.13]

13. Secondary Outcome: Partial Metabolic Response (PMR), Cycle 1
Description: Partial metabolic responses measured by 2-[F-18]-fluoro-2-deoxy-D-glucose positron emission tomography (FDG-PET) (or FDG-PET/Computed Tomography (CT)) with a comparison to baseline (pre-dose)
Time Frame: Cycle 1 Day 8
Population: Efficacy analysis set
Measure: Number; unit: Participants
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 6 | 8 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |

14. Secondary Outcome: Partial Metabolic Response (PMR), Cycle 2
Description: as for outcome 13
Time Frame: Cycle 2 Day 8
Population: Efficacy analysis set
Measure: Number; unit: Participants
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 6 | 8 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 5 |  |  |  |  |  |  |  |  |  |  |  |  |  |

15. Secondary Outcome: Complete Metabolic Response (CMR), Cycle 1
Description: Complete metabolic responses measured by 2-[F-18]-fluoro-2-deoxy-D-glucose positron emission tomography (FDG-PET) (or FDG-PET/Computed Tomography (CT)) with a comparison to baseline (pre-dose)
Time Frame: Cycle 1 Day 8
Population: Efficacy analysis set
Measure: Number; unit: Participants
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 6 | 8 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |

16. Secondary Outcome: Complete Metabolic Response (CMR), Cycle 2
Description: as for outcome 15
Time Frame: Cycle 2 Day 8
Population: Efficacy analysis set
Measure: Number; unit: Participants
Arm/Group | Part A 25mg BD Soln Cont | Part A 50mg BD Soln Cont | Part B 50mg BD Soln Cont | Part B Fed/Fasted 50mg BD Tab Cont | Part A 75mg QD Soln Cont | Part A 125mg QD Soln Cont | Part A 100mg QD Tab Cont | Part A 125mg QD Tab Cont | Part A 175mg QD Tab Cont | Part A 100mg BD Tab Int | Part A 125mg BD Tab Int | Part A 170mg BD Tab Int | Part A 225mg BD Tab Int | Part B 125mg BD Tab Int | Part B 170mg BD Tab Int | Part A 70mg BD Soln Cont | Part A 100mg BD Soln Cont
Number analyzed (Participants) | 6 | 8 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: At each visit from screening through to 30 day follow up (estimated to be up to 4 months, plus 30 days follow up)
Description: Continuous BD solution dosing cohorts 25mg, 50mg, 70mg, 100mg Continuous BD tablet dosing cohort Fed/Fasted 50mg Continuous QD solution dosing cohorts 75mg, 125mg Continuous Qd tablet dosing cohorts 100mg, 125mg, 175mg Intermmittent BD tablet dosing cohorts 100mg, 125mg, 170mg, 225mg
Groups:
- Part A - AZD2014 100 mg BD Solution; Part A - AZD2014 25 mg BD Solution; Part A - AZD2014 50 mg BD Solution; Part A - AZD2014 70 mg BD Solution; Part B - AZD2014 50 mg BD Solution; Part B - AZD2014 50 mg BD Tablet Fasted/Fed; Part B - AZD2014 BD 50 mg Tablet Fed/Fasted: Continuous BD dosing
- Part A - AZD2014 100 mg QD Tablet; Part A - AZD2014 125 mg QD Tablet; Part A - AZD2014 175 mg QD Tablet; Part A - AZD2014 75 mg QD Solution: Continuous QD dosing
- Part A - AZD2014 125 mg QD Solution: Continous QD dosing
- Part A - Intermittent AZD2014 100 mg BD Tablet; Part A - Intermittent AZD2014 125 mg BD Tablet; Part A - Intermittent AZD2014 170 mg BD Tablet; Part A - Intermittent AZD2014 225 mg BD Tablet; Part B - Intermittent AZD2014 125 mg BD Tablet; Part B - Intermittent AZD2014 170 mg BD Tablet: Intermittent BD dosing
Arm/Group | Part A - AZD2014 100 mg BD Solution | Part A - AZD2014 100 mg QD Tablet | Part A - AZD2014 125 mg QD Solution | Part A - AZD2014 125 mg QD Tablet | Part A - AZD2014 175 mg QD Tablet | Part A - AZD2014 25 mg BD Solution | Part A - AZD2014 50 mg BD Solution | Part A - AZD2014 70 mg BD Solution | Part A - AZD2014 75 mg QD Solution | Part A - Intermittent AZD2014 100 mg BD Tablet | Part A - Intermittent AZD2014 125 mg BD Tablet | Part A - Intermittent AZD2014 170 mg BD Tablet | Part A - Intermittent AZD2014 225 mg BD Tablet | Part B - AZD2014 50 mg BD Solution | Part B - AZD2014 50 mg BD Tablet Fasted/Fed | Part B - AZD2014 BD 50 mg Tablet Fed/Fasted | Part B - Intermittent AZD2014 125 mg BD Tablet | Part B - Intermittent AZD2014 170 mg BD Tablet
Serious Adverse Events (participants affected / at risk) | 1/4 | 4/8 | 0/5 | 2/3 | 4/7 | 5/6 | 0/8 | 2/5 | 1/3 | 1/3 | 3/7 | 3/8 | 6/8 | 11/33 | 4/9 | 3/9 | 3/6 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 8/8 | 5/5 | 3/3 | 7/7 | 6/6 | 8/8 | 5/5 | 3/3 | 3/3 | 7/7 | 8/8 | 8/8 | 32/33 | 9/9 | 9/9 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - AZD2014 100 mg BD Solution (N=4) | Part A - AZD2014 100 mg QD Tablet (N=8) | Part A - AZD2014 125 mg QD Solution (N=5) | Part A - AZD2014 125 mg QD Tablet (N=3) | Part A - AZD2014 175 mg QD Tablet (N=7) | Part A - AZD2014 25 mg BD Solution (N=6) | Part A - AZD2014 50 mg BD Solution (N=8) | Part A - AZD2014 70 mg BD Solution (N=5) | Part A - AZD2014 75 mg QD Solution (N=3) | Part A - Intermittent AZD2014 100 mg BD Tablet (N=3) | Part A - Intermittent AZD2014 125 mg BD Tablet (N=7) | Part A - Intermittent AZD2014 170 mg BD Tablet (N=8) | Part A - Intermittent AZD2014 225 mg BD Tablet (N=8) | Part B - AZD2014 50 mg BD Solution (N=33) | Part B - AZD2014 50 mg BD Tablet Fasted/Fed (N=9) | Part B - AZD2014 BD 50 mg Tablet Fed/Fasted (N=9) | Part B - Intermittent AZD2014 125 mg BD Tablet (N=6) | Part B - Intermittent AZD2014 170 mg BD Tablet (N=3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - AZD2014 100 mg BD Solution (N=4) | Part A - AZD2014 100 mg QD Tablet (N=8) | Part A - AZD2014 125 mg QD Solution (N=5) | Part A - AZD2014 125 mg QD Tablet (N=3) | Part A - AZD2014 175 mg QD Tablet (N=7) | Part A - AZD2014 25 mg BD Solution (N=6) | Part A - AZD2014 50 mg BD Solution (N=8) | Part A - AZD2014 70 mg BD Solution (N=5) | Part A - AZD2014 75 mg QD Solution (N=3) | Part A - Intermittent AZD2014 100 mg BD Tablet (N=3) | Part A - Intermittent AZD2014 125 mg BD Tablet (N=7) | Part A - Intermittent AZD2014 170 mg BD Tablet (N=8) | Part A - Intermittent AZD2014 225 mg BD Tablet (N=8) | Part B - AZD2014 50 mg BD Solution (N=33) | Part B - AZD2014 50 mg BD Tablet Fasted/Fed (N=9) | Part B - AZD2014 BD 50 mg Tablet Fed/Fasted (N=9) | Part B - Intermittent AZD2014 125 mg BD Tablet (N=6) | Part B - Intermittent AZD2014 170 mg BD Tablet (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 2 (4) | 6 (7) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Halo vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (3) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 2 (2) | 3 (4) | 2 (2) | 3 (4) | 10 (15) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 2 (3) | 2 (2) | 4 (7) | 2 (3) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 4 (7) | 3 (5) | 16 (23) | 4 (4) | 3 (3) | 3 (4) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 5 (14) | 4 (4) | 1 (2) | 5 (6) | 2 (2) | 3 (4) | 3 (3) | 2 (4) | 1 (1) | 4 (6) | 7 (11) | 6 (9) | 16 (23) | 3 (4) | 4 (5) | 4 (4) | 2 (2)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (4) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 8 (9) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (4) | 5 (6) | 3 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (12) | 5 (8) | 10 (15) | 2 (3) | 3 (4) | 2 (4) | 1 (1)
Application site vesicles (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 7 (8) | 4 (5) | 2 (3) | 3 (4) | 2 (2) | 5 (5) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 5 (6) | 4 (6) | 23 (23) | 5 (6) | 3 (3) | 5 (5) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (4) | 1 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (5) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Heart rate abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary physical examination abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field tests (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5) | 3 (4) | 4 (4) | 2 (3) | 5 (5) | 3 (3) | 5 (6) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 4 (5) | 12 (14) | 4 (5) | 4 (5) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 4 (5) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 4 (10) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 6 (7) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 8 (8) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (10) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 10 (16) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less